CLINICAL TRIAL: NCT05021705
Title: Non Diabetic Causes of Chronic Kidney Disease in Type 2 Diabetic Patients
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Asmaa Nady Sayed, principal investigator, Assiut University
Other Study IDs: Non diabetic kidney disease
Record Dates: First submitted 2021-08-19; First posted 2021-08-25 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Diabetic Kidney Disease
MeSH Terms: conditions — Diabetic Nephropathies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Determination of the possible causes of chronic kidney disease (CKD) in patients with type 2 diabetes mellitus with an atypical presentations of renal disease for proper management and thus improving renal outcome.

DETAILED DESCRIPTION:
Diabetes mellitus (DM) is one of the most important health problems worldwide, and its prevalence is increasing. One of the complications of DM is diabetic kidney disease (DKD), which is responsible for over 40% of cases of chronic kidney disease requiring dialysis or kidney transplantation in the Western world.

The natural history of DKD in patients with type 1 DM is well characterized because we know the precise time of DM onset. Classically, these patients develop microalbuminuria, followed by macroalbuminuria in the first 15 years of DM. After 20 years of DM, progressive loss of glomerular filtration rate (GFR) develops. The majority of these patients have diabetic retinopathy. However, the natural history of renal disease in adults with DM type 2 is controversial. Before diagnosis, type 2 DM has usually evolved over several years but has remained unnoticed.

In 2007, KDOQI guidelines described characteristics of diabetic patients that indicate DKD involvement, namely the presence of macroalbuminuria or microalbuminuria with diabetic retinopathy in both types of DM, and in type 1 DM patients, over 10 years of DM. In addition, the guidelines summarize the characteristics that suggest the presence of non-diabetic kidney disease (NDKD): absence of diabetic retinopathy, fast decline of renal function, fast increase in proteinuria or nephrotic syndrome, refractory hypertension, active urinary sediment or signs or symptoms of systemic disease or>30% reduction in GFR within 2-3 months after starting the blockade of the renin-angiotensin-aldosterone system (RAAS).Yuan 2017 addressed the accuracy of a clinical diagnosis of DKD among diabetic patients following the criteria proposed by the KDOQI guidelines. Around 20% of patients did not meet KDOQI criteria for DKD in type 2 DM, suggesting a significant over estimation of DKD in this population. This high proportion of NDKD matches previous publications which demonstrated that about a third of patients with DM have biopsy-proven NDKD. The gold standard for diagnosis is renal biopsy. Renal biopsy in diabetic patients has focused on identifying NDKD, because these patients have different prognosis and therapy. The most frequent biopsy indications in diabetic patients are nephrotic syndrome, nephrotic proteinuria in patients with < 5 years of DKD evolution, microhaematuria, acute kidney injury and unexplained decline of renal function. Several groups have studied renal biopsies from diabetic patients, showing that the most frequent NDKD diagnoses are IgA nephropathy, membranous nephropathy and focal segmental glomerulosclerosis.

Different studies have shown that patients with DKD have a worse renal prognosis and that the prevalence of NDKD is high in diabetic patients. Therefore, it is important to accurately classify diabetic patients for DKD or NDKD. Yuan 2017 studied the differential characteristics between patients meeting clinical criteria to diagnose DKD according to KDOQI and misclassified patients. They showed that those patients lacking KDOQI-predicted DKD were more likely to have an active urine sediment and less likely to have developed macroalbuminuria or retinopathy prior to end-stage renal disease. Using the logistic regression analysis, diabetic retinopathy was the only factor independently associated with patients who met KDOQI criteria.

Kidney biopsy studies in diabetic patients have found predictive factors for NDKD: absence of diabetic retinopathy, low glycosylated haemoglobin, worse renal function, lower level of proteinuria, the presence of microscopic haematuria, older age and shorter DM evolution. Although the Yuan 2017 cohort is small and the diagnostic method was usually not renal biopsy, the results are in line with prior reports. However, recent studies have shown that patients with biopsy-proven DKD may be normoalbuminuric. Thus, further studies with larger cohorts and ideally renal biopsy confirmation are necessary to find factors better predicting NDKD in type 2 diabetic patients. These studies may help to design novel diagnostic tools to be applied by physicians in daily clinical practice. New therapeutic agents for the treatment of DKD have recently been characterized. Endothelin receptor antagonists, sodium glucose co-transporter2 inhibitors, incretins and agents targeting inflammation/fibrosis are probably the most promising candidates on top of the classical RAAS blockers. Therefore, it is mandatory that patients with diabetic renal disease are adequately classified, differentiating clearly those with DKD and those with NDKD. In addition, among those with DKD, a reliable classification within different pathological categories will be of great value to individualize treatment strategies.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes mellitus having proteinuria associated with macroscopic or microscopic haematuria.
* Patients with type 2 diabetes mellitus with nephrotic syndrome appearing in the early stages of DM (less than 10 years of diagnosis) in absence of retinopathy or neuropathy.
* Patients with type 2 diabetes mellitus with unexplained renal failure or rapidly progressive renal dysfunction within few weeks or months.
* Patients with type 2 diabetes mellitus with symptoms and signs suggestive of systemic disease that may affect the kidney as SLE, vasculitis, multiple myeloma or lymphoma.
* Patients with type 2 diabetes mellitus with rapidly progressive glomerulonephritis.

Exclusion Criteria:

* Patients with type 1 diabetes mellitus.
* DM with clinically, laboratory or radiologically evident CKD due to either chronic pyelonephritis, polycystic kidney disease or chronic obstructive nephropathy.
* DM with end stage renal disease (ESRD) with bilateral small kidneys.
* Patients with any contraindication to renal biopsy (systemic infections, bleeding tendency, low platelets, decrease prothrombin concentration).

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Type 2 Diabetic patients
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2020-05 (Actual)

PRIMARY OUTCOMES:
renal biopsy | baseline
  The preferred site for renal biopsy was the lateral aspect of the lower pole of the left kidney under ultrasound guidance with the patient in the prone position and local anesthesia was used. An automated biopsy gun and a 16 gauge needle was used to ensure the biopsy sample contained a minimum of ten glomeruli. After biopsy compression on site of biopsy was done and strict follow up for the patient to exclude any complications. No complications were occurred for any patients. Renal biopsy specimens were prepared according to standard methods for light microscopy and immunoperoxidase. Electron microscopy was not routinely performed.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Espinel E, Agraz I, Ibernon M, Ramos N, Fort J, Seron D. Renal Biopsy in Type 2 Diabetic Patients. J Clin Med. 2015 May 18;4(5):998-1009. doi: 10.3390/jcm4050998. PMID 26239461
- [Background] Kramer A, Pippias M, Noordzij M, Stel VS, Afentakis N, Ambuhl PM, Andrusev AM, Fuster EA, Arribas Monzon FE, Asberg A, Barbullushi M, Bonthuis M, Caskey FJ, Castro de la Nuez P, Cernevskis H, des Grottes JM, Garneata L, Golan E, Hemmelder MH, Ioannou K, Jarraya F, Kolesnyk M, Komissarov K, Lassalle M, Macario F, Mahillo-Duran B, Martin de Francisco AL, Palsson R, Pechter U, Resic H, Rutkowski B, Santiuste de Pablos C, Seyahi N, Simic Ogrizovic S, Slon Roblero MF, Spustova V, Stojceva-Taneva O, Traynor J, Massy ZA, Jager KJ. The European Renal Association - European Dialysis and Transplant Association (ERA-EDTA) Registry Annual Report 2015: a summary. Clin Kidney J. 2018 Feb;11(1):108-122. doi: 10.1093/ckj/sfx149. Epub 2018 Jan 5. PMID 29423210
- [Background] Lytvyn Y, Bjornstad P, Pun N, Cherney DZ. New and old agents in the management of diabetic nephropathy. Curr Opin Nephrol Hypertens. 2016 May;25(3):232-9. doi: 10.1097/MNH.0000000000000214. PMID 26890303
- [Background] Kramer HJ, Nguyen QD, Curhan G, Hsu CY. Renal insufficiency in the absence of albuminuria and retinopathy among adults with type 2 diabetes mellitus. JAMA. 2003 Jun 25;289(24):3273-7. doi: 10.1001/jama.289.24.3273. PMID 12824208
- [Background] KDOQI. KDOQI Clinical Practice Guidelines and Clinical Practice Recommendations for Diabetes and Chronic Kidney Disease. Am J Kidney Dis. 2007 Feb;49(2 Suppl 2):S12-154. doi: 10.1053/j.ajkd.2006.12.005. No abstract available. PMID 17276798
- [Background] Yuan CM, Nee R, Ceckowski KA, Knight KR, Abbott KC. Diabetic nephropathy as the cause of end-stage kidney disease reported on the medical evidence form CMS2728 at a single center. Clin Kidney J. 2017 Apr;10(2):257-262. doi: 10.1093/ckj/sfw112. Epub 2016 Dec 22. PMID 28396744
- [Background] Bermejo S, Soler MJ, Gimeno J, Barrios C, Rodriguez E, Mojal S, Pascual J. Predictive factors for non-diabetic nephropathy in diabetic patients. The utility of renal biopsy. Nefrologia. 2016 Sep-Oct;36(5):535-544. doi: 10.1016/j.nefro.2016.06.006. Epub 2016 Aug 11. English, Spanish. PMID 27523263
- [Background] Fiorentino M, Bolignano D, Tesar V, Pisano A, Van Biesen W, D'Arrigo G, Tripepi G, Gesualdo L; ERA-EDTA Immunonephrology Working Group. Renal Biopsy in 2015--From Epidemiology to Evidence-Based Indications. Am J Nephrol. 2016;43(1):1-19. doi: 10.1159/000444026. Epub 2016 Feb 5. PMID 26844777
- [Background] Sharma SG, Bomback AS, Radhakrishnan J, Herlitz LC, Stokes MB, Markowitz GS, D'Agati VD. The modern spectrum of renal biopsy findings in patients with diabetes. Clin J Am Soc Nephrol. 2013 Oct;8(10):1718-24. doi: 10.2215/CJN.02510213. Epub 2013 Jul 25. PMID 23886566
- [Background] Bi H, Chen N, Ling G, Yuan S, Huang G, Liu R. Nondiabetic renal disease in type 2 diabetic patients: a review of our experience in 220 cases. Ren Fail. 2011;33(1):26-30. doi: 10.3109/0886022X.2010.536292. PMID 21219202
- [Background] Byun JM, Lee CH, Lee SR, Moon JY, Lee SH, Lee TW, Ihm CG, Jeong KH. Renal outcomes and clinical course of nondiabetic renal diseases in patients with type 2 diabetes. Korean J Intern Med. 2013 Sep;28(5):565-72. doi: 10.3904/kjim.2013.28.5.565. Epub 2013 Aug 14. PMID 24009452
- [Background] Chong YB, Keng TC, Tan LP, Ng KP, Kong WY, Wong CM, Cheah PL, Looi LM, Tan SY. Clinical predictors of non-diabetic renal disease and role of renal biopsy in diabetic patients with renal involvement: a single centre review. Ren Fail. 2012;34(3):323-8. doi: 10.3109/0886022X.2011.647302. Epub 2012 Jan 17. PMID 22250665
- [Background] Liu MY, Chen XM, Sun XF, Zhou JH, Zhang XG, Zhu HY, Chen YZ, Liu SW, Wei RB, Tang L, Cai GY, Zhang L, Bai XY. Validation of a differential diagnostic model of diabetic nephropathy and non-diabetic renal diseases and the establishment of a new diagnostic model. J Diabetes. 2014 Nov;6(6):519-26. doi: 10.1111/1753-0407.12150. Epub 2014 Apr 25. PMID 24645648
- [Background] Wilfred DC, Mysorekar VV, Venkataramana RS, Eshwarappa M, Subramanyan R. Nondiabetic Renal Disease in type 2 Diabetes Mellitus Patients: A Clinicopathological Study. J Lab Physicians. 2013 Jul;5(2):94-9. doi: 10.4103/0974-2727.119850. PMID 24701101
- [Background] Chang TI, Park JT, Kim JK, Kim SJ, Oh HJ, Yoo DE, Han SH, Yoo TH, Kang SW. Renal outcomes in patients with type 2 diabetes with or without coexisting non-diabetic renal disease. Diabetes Res Clin Pract. 2011 May;92(2):198-204. doi: 10.1016/j.diabres.2011.01.017. Epub 2011 Feb 12. PMID 21320734
- [Background] Wong TY, Choi PC, Szeto CC, To KF, Tang NL, Chan AW, Li PK, Lai FM. Renal outcome in type 2 diabetic patients with or without coexisting nondiabetic nephropathies. Diabetes Care. 2002 May;25(5):900-5. doi: 10.2337/diacare.25.5.900. PMID 11978688
- [Background] Soleymanian T, Hamid G, Arefi M, Najafi I, Ganji MR, Amini M, Hakemi M, Tehrani MR, Larijani B. Non-diabetic renal disease with or without diabetic nephropathy in type 2 diabetes: clinical predictors and outcome. Ren Fail. 2015 May;37(4):572-5. doi: 10.3109/0886022X.2015.1007804. Epub 2015 Feb 16. PMID 25682971
- [Background] Robles NR, Villa J, Gallego RH. Non-Proteinuric Diabetic Nephropathy. J Clin Med. 2015 Sep 7;4(9):1761-73. doi: 10.3390/jcm4091761. PMID 26371050
- [Background] Anguiano L, Riera M, Pascual J, Soler MJ. Endothelin Blockade in Diabetic Kidney Disease. J Clin Med. 2015 May 25;4(6):1171-92. doi: 10.3390/jcm4061171. PMID 26239552
- [Background] Fioretto P, Mauer M. Histopathology of diabetic nephropathy. Semin Nephrol. 2007 Mar;27(2):195-207. doi: 10.1016/j.semnephrol.2007.01.012. PMID 17418688
- [Background] Tervaert TW, Mooyaart AL, Amann K, Cohen AH, Cook HT, Drachenberg CB, Ferrario F, Fogo AB, Haas M, de Heer E, Joh K, Noel LH, Radhakrishnan J, Seshan SV, Bajema IM, Bruijn JA; Renal Pathology Society. Pathologic classification of diabetic nephropathy. J Am Soc Nephrol. 2010 Apr;21(4):556-63. doi: 10.1681/ASN.2010010010. Epub 2010 Feb 18. PMID 20167701